CLINICAL TRIAL: NCT04281433
Title: Electromicrographic Activity as Well as Clinical Performance of Bulk Fill Composite With Activa Bioactive Liner
Brief Title: Clinical Performance of Bulk Fill Composite With Activa Bioactive Liner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim Ahmed, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC16-051
Record Dates: First submitted 2020-02-11; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Clinical Study of Activa Bioactive Restorative; Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- unilateral (Experimental)
  Interventions: Other: Activa Bioactive
- bilateral (Experimental)
  Interventions: Other: Activa Bioactive

INTERVENTIONS:
Other: Activa Bioactive — Before cavity preparation and restoration, masticatory muscles activity will be evaluated by using electromyography. An electromyography detects the electrical potential generated by muscle cells. A total of 40 posterior teeth will be selected for this study and grouped into 2 main groups (20 for each group)) according to presence of caries in one or both side in patient (unilateral or bilateral). Split mouth technique will be used. The affected teeth will be treated by removing the caries and restored tooth with bulk fill composite material, after restoring the affected teeth. Masticatory muscles activity will be evaluated by using electromyography to detect any changes in masticatory muscles activity before and after restoration.

SUMMARY:
electromyographic activity as well as clinical performance of bulk-Fill composite resins with Activa Bioactive Liner

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-40 years and cooperative patient.
* Good oral hygiene.
* Normal occlusal relation with normal dentition.

Exclusion Criteria:

* Patient with severe medical problems.
* Tenderness with percussion or pre-operative pulpal pain.
* Mobile tooth and tooth with gingival recession.
* Pregnant or lactating females.
* Cracked teeth or teeth with deep periodontal pockets.
* Tooth with previous restoration.
* Allergy to resin materials.
* Defective restorations adjacent or opposing to tooth.
* Patient with bruxism

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Electromyographic activity | baseline (immediate)
  An electromyography detects the electrical potential generated by muscle cells. When these cells are electrically activated, the signals can be analyzed to detect medical Abnormalities, activation level, or recruitment order, or to analyze the biomechanics of human movement
Electromyographic activity | one week
  An electromyography detects the electrical potential generated by muscle cells. When these cells are electrically activated, the signals can be analyzed to detect medical Abnormalities, activation level, or recruitment order, or to analyze the biomechanics of human movement
Electromyographic activity | after three months
  An electromyography detects the electrical potential generated by muscle cells. When these cells are electrically activated, the signals can be analyzed to detect medical Abnormalities, activation level, or recruitment order, or to analyze the biomechanics of human movement
Electromyographic activity | after six months
  An electromyography detects the electrical potential generated by muscle cells. When these cells are electrically activated, the signals can be analyzed to detect medical Abnormalities, activation level, or recruitment order, or to analyze the biomechanics of human movement

SECONDARY OUTCOMES:
Survival rate of restorative material | six months
  USPHS criteria

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar University, Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided